CLINICAL TRIAL: NCT00941941
Title: Comparison of Non-mesh (Desarda) and Mesh (Lichtenstein) Methods for Inguinal Hernia Repair at Mulago Hospital: a Double-blind Randomised Controlled Trial
Brief Title: Non-Mesh Versus Mesh Method for Inguinal Hernia Repair
Acronym: IHR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Makerere University (Other)
Collaborators: Mulago Hospital, Uganda (Other)
Responsible Party: William Manyilirah, Makerere University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2006/HD11/6219U; REC REF 2009-080
Record Dates: First submitted 2009-07-11; First posted 2009-07-20 (Estimated); Last update posted 2009-07-20 (Estimated); Status verified 2009-07

CONDITIONS: Hernia, Inguinal
Keywords: Inguinal; Hernia; Hernia-repair; Non-mesh; Mesh; Desarda; Lichtenstein
MeSH Terms: conditions — Hernia, Inguinal; Hernia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Non-mesh Hernia Repair (Experimental): Reinforcement with a strip of external oblique aponeurosis
  Interventions: Procedure: Non-mesh Hernia Repair
- Mesh Hernia Repair (Active Comparator): Polypropylene mesh placement
  Interventions: Procedure: Mesh Hernia Repair

INTERVENTIONS:
Procedure: Non-mesh Hernia Repair — Non-mesh method for treatment of inguinal hernia without the use of a foreign material (mesh). It involves reinforcement of the weakened posterior wall of inguinal canal with a small, undetached strip of aponeurotic tissue of external
  Other Names: Desarda repair
  Arms: Non-mesh Hernia Repair
Procedure: Mesh Hernia Repair — Mesh method for treatment of inguinal hernias by use of an implant (mesh) to reinforce the weakened posterior wall of the inguinal canal. The mesh is made of polypropylene material.
  Other Names: Lichtenstein repair
  Arms: Mesh Hernia Repair

SUMMARY:
The study aims at establishing the effectiveness of the non-mesh (Desarda) technique for the treatment of primary inguinal hernias at Mulago Hospital in Uganda. First developed and used in India, the Desarda method is reported to offer superior outcomes such as minimal postoperative groin pain and near zero recurrence rates. In comparison to the mesh-based repairs, it is a simple and affordable technique suitable for the resource-constrained communities. It is devoid of complications associated with foreign body implants. Early clinical outcomes which include acute groin pain, time to resumption of normal gait, operative time and complications will be assessed. Participants will be followed at 2 hours, 3 days, 7 days and 14 days postoperatively.

The investigators hypothesize that the mean postoperative acute groin pain score, or the mean postoperative day of return to normal gait is different in adult patients who undergo the non-mesh (Desarda) repair from what it is in those who undergo the mesh (Lichtenstein) technique of hernia repair.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 and above;
* with a primary, reducible inguinal or inguino-scrotal hernia;
* who consent to participate in the study;
* who have a telephone contact.

Exclusion Criteria:

* Giant inguino-scrotal hernias;
* Obstructive uropathy or chronic obstructive pulmonary disease;
* Impaired mental state and are unable to give an accurate assessment of the key outcomes of the operation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2009-05; Primary Completion 2009-08 (Estimated); Study Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
Acute groin pain after surgery (measured on pain visual analogue scale of 0-10) | 2 Weeks
Time (in days) taken to return to normal gait | 2 Weeks

SECONDARY OUTCOMES:
Operative time (in Minutes) | 2 hours
Complications during and after surgery | 2 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: William Manyilirah, Principal Investigator — Makerere University; Alex Upoki, Study Chair — Makerere University
Locations (1):
- Mulago National Referral Hospital, Kampala, Central Region, Uganda